CLINICAL TRIAL: NCT04072055
Title: MOTO MEDIAL UNICOMPARTMENTAL KNEE ARTHROPLASTY: OPEN, PROSPECTIVE, MULTICENTRIC, OBSERVATIONAL STUDY
Brief Title: MOTO Post-marketing Surveillance Study
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulty in the centers
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.021.01
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Osteonecrosis; Osteo Arthritis Knee
Keywords: Unicompartmental Knee Arthroplasty; UKA; antomic femoral component; anatomic tibial component
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MOTO medial: Patients suitable fulfilling the standard criteria for the implantation of unicondylar implant.
  Interventions: Device: MOTO Medial

INTERVENTIONS:
Device: MOTO Medial — MOTO medial unicompartmental knee system

SUMMARY:
The prospective, multicentric, observational study has the aims to monitor the performance of the MOTO medial unicompartmental knee system in the treatment of patients with knee disease requiring a UKA. 150 patients will be recruited in 18 months and will be reviewed until 5 years follow-up visit after surgery. The primary objective of the study is to evaluate the prosthesis survival at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unicompartmental tibiofemoral osteoarthritis (OA) of the knee that meet the indications for use of Medacta implant included in this study (on-label use);
* Patients suffering from unilateral osteoarthritis or osteonecrosis of a single knee compartment;
* Frontal deformity < 10° (evaluated on weight-bearing long-axis x-rays);
* Flexion contracture < 10°;
* Intact ligaments;
* Patients willing and able to provide written informed consent for participation in the study;
* Patient's age over 18 years old;
* Patient with BMI < 40 kg/m2;
* Patients willing to comply with the pre and post-operative evaluation schedule.

Exclusion Criteria:

* Patients with one or more medical conditions identified as a contraindication in the labelling on any Medacta implants used in this study;
* Any patient who cannot or will not provide informed consent for participation in the study;
* Patients who need a revision surgery;
* Patients who had previously undergone high tibial osteotomy or anterior cruciate ligament (ACL) reconstruction;
* Patients with BMI ≥ 40 kg/m2;
* Patients unable to understand and take action;
* Any case not described in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Prosthesis survival | 5 years
  survivorship analysis according to Kaplan-Meier method at 5 years after surgery

SECONDARY OUTCOMES:
New Knee Society Score (KSS) | preoperative, 3 months, 1, 3 and 5 years
  Functionality and symptom of operated knee will be evaluated by New KSS score
Radiological analysis | preoperative, postoperative, 3 months, 1, 3 and 5 years
  Postoperative stability and fixation of the device will be assessed by standard radiological exams
Complication | up to 5 years
  Intraoperative and postoperative complication will be collected during all duration of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Zeno Campus Knokke-Heist, Knokke-Heist
  - Clinique Saint-Joseph, Liège

IPD SHARING:
Plan to Share IPD: Undecided